CLINICAL TRIAL: NCT06167642
Title: Assessing the Modulation of Retinal Atrophy and Neurofilament Light Chain by Ofatumumab in Relapsing Multiple Sclerosis
Brief Title: Retinal Atrophy and Neurofilament Light Chain in People With Multiple Sclerosis Taking Ofatumumab
Status: Enrolling by invitation | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00347678
Record Dates: First submitted 2023-11-15; First posted 2023-12-12 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis; Tomography, Optical Coherence; Retinal Degeneration; Visual Acuity
MeSH Terms: conditions — Multiple Sclerosis; Retinal Degeneration | interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- People with RMS due to commence or already receiving ofatumumab therapy: 75 people with RMS due to commence or already receiving ofatumumab therapy within 60 days of baseline.
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — Ofatumumab therapy is part of the patient's clinical care and is not given as part of the study
  Other Names: Kesimpta

SUMMARY:
This study aims to assess whether, and the degree to which, ofatumumab modulates or reduces rates of retinal atrophy in people with relapsing-remitting MS (RMS), according to baseline serum neurofilament light chain (sNfL) levels.

DETAILED DESCRIPTION:
Seventy-five people with RMS who due to commence or already receiving ofatumumab therapy within 60 days of baseline will be recruited. All recruited participants will be tracked prospectively over a two-year period. Participants will complete an optical coherence tomography (OCT) scan, visual acuity (VA) assessments, EDSS, and sNfL blood level at baseline and every 6 months. Participants will be tracked prospectively for 2 years. OCT scans, sNfL levels, disability score determinations, 100% high-contrast, 2.5% and 1.25% low-contrast letter acuities will be performed every 6 months. Results from an existing cohort of approximately 75 healthy controls (HC) from a separate study undergoing annual OCT and visual function assessments will be used for comparison purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 - 70 years of age
2. Have RMS as confirmed by the treating neurologist based on the 2017 revised McDonald criteria

   AND Either
   * be due to commence ofatumumab within 60 days of baseline OCT/VA/phlebotomy or
   * be existing patients attending the center and already receiving ofatumumab, be eligible for inclusion, and already undergoing all of the proposed study procedures.
3. Willing to sign informed consent
4. Willing to undergo phlebotomy

Exclusion Criteria:

* Uncontrolled Diabetes
* Uncontrolled Hypertension
* Glaucoma
* Refractive errors of +/- 6 diopters
* Other neurologic or ophthalmologic disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 75 people with RMS due to commence or already receiving ofatumumab therapy within 60 days of baseline OCT, VA, and blood draw.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Ganglion cell inner plexiform (GCIP) atrophy in RMS relative to HCs, according to baseline sNfL levels | at least 12 months for up to 2 years
  Rates of of GCIP layer thinning (µm/year) will be assessed according to baseline sNfL levels using mixed-effects linear regression models with random subject and eye-specific random intercepts and random slopes in time, using time from baseline OCT visit (in years) as a continuous variable in both unadjusted models (including time, sNfL group and their interaction) and models adjusted for the cross-sectional and longitudinal effects of covariates (age, sex, race, and history of optic neuritis) by including these variables and their respective interactions with time.

SECONDARY OUTCOMES:
Inner nuclear layer (INL) atrophy in RMS relative to HCs | at least 12 months for up to 2 years
  Rates of INL layer thinning (µm/year) will be assessed according to baseline sNfL levels using mixed-effects linear regression models with random subject and eye-specific random intercepts and random slopes in time, using time from baseline OCT visit (in years) as a continuous variable in both unadjusted models (including time, sNfL group and their interaction) and models adjusted for the cross-sectional and longitudinal effects of covariates (age, sex, race, and history of optic neuritis) by including these variables and their respective interactions with time.
Outer nuclear layer (ONL) atrophy in RMS relative to HCs | at least 12 months for up to 2 years
  Rates of INL and ONL layer thinning (µm/year) will be assessed according to baseline sNfL levels using mixed-effects linear regression models with random subject and eye-specific random intercepts and random slopes in time, using time from baseline OCT visit (in years) as a continuous variable in both unadjusted models (including time, sNfL group and their interaction) and models adjusted for the cross-sectional and longitudinal effects of covariates (age, sex, race, and history of optic neuritis) by including these variables and their respective interactions with time.
Differences in the visual function scores | at least 12 months for up to 2 years
  Exploratory analyses within the ofatumumab group will assess changes in visual function scores by baseline sNfL levels utilizing logistic regression.
Differences in expanded disability status scale (EDSS) scores | at least 12 months for up to 2 years
  Exploratory analyses within the ofatumumab group will assess changes in EDSS scores by baseline sNfL levels utilizing logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Shiv Saidha, MBBCh, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States